CLINICAL TRIAL: NCT04943497
Title: A Prospective Observational Study to Describe Clinical Outcomes, Treatment Patterns, Patients Characteristics Among Patients With HR+/HER2- Advanced BC Initiating Treatment With Risarg® (Ribociclib), Piqray® (Alpelisib), Endocrine Therapy or Chemotherapy in Routine Clinical Practice in Russia
Brief Title: A Prospective Observational Study to Describe Clinical Outcomes, Treatment Patterns, Patients Characteristics Among Patients With HR+/HER2- Advanced BC Initiating Treatment With Risarg®, Piqray®, Endocrine Therapy or Chemotherapy in Routine Clinical Practice in Russia
Acronym: PROSPERITY
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011ARU01
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; CDK4/6 inhibitors; advanced HR+/HER2- breast cancer; ribociclib; Risarg; alpelisib; Piqray; Russia
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- ribociclib + AI/fulvestrant: Patients administered ribociclib + AI/fulvestrant by prescription AI: Aromatase inhibitor
  Interventions: Other: ribociclib
- aplelicib + fulvestrant: Patients administered aplelicib + fulvestrant by prescription
  Interventions: Other: aplelicib
- mono endocrine therapy: Patients administered mono endocrine therapy by prescription
  Interventions: Other: mono endocrine therapy
- chemotherapy: Patients administered chemotherapy by prescription
  Interventions: Other: chemotherapy

INTERVENTIONS:
Other: ribociclib — There is no treatment allocation. Patients administered ribociclib by prescription that have started before inclusion of the patient into the study will be enrolled.
  Groups: ribociclib + AI/fulvestrant
Other: aplelicib — There is no treatment allocation. Patients administered aplelicib by prescription that have started before inclusion of the patient into the study will be enrolled.
  Groups: aplelicib + fulvestrant
Other: mono endocrine therapy — There is no treatment allocation. Patients administered mono endocrine therapy by prescription that have started before inclusion of the patient into the study will be enrolled.
  Groups: mono endocrine therapy
Other: chemotherapy — There is no treatment allocation. Patients administered chemotherapy by prescription that have started before inclusion of the patient into the study will be enrolled.
  Groups: chemotherapy

SUMMARY:
This study is planned as a prospective multicenter NIS. This study is observational in nature and does not impose a therapy protocol, diagnostic/therapeutic interventions or a visit schedule. Patients with HR+/ HER2- advanced or metastatic BC that initiated treatment with ribociclib, alpelisib, mono endocrine therapy or chemotherapy will be included into the study across seven Russian districts.

DETAILED DESCRIPTION:
Patients will attend the sites in accordance with routine clinical practice. It is assumed that visits will be conducted every 3-4 months. Patients will undergo standard procedures and tests according to clinical guidelines and physician's judgement. Available data from routine clinical management of the patients will be collected at patients' visits to the clinical site. Patients enrolled in the study will be followed up until death or study close whichever occurs first. The recruitment period is planned for 24 months, observation period for maximum of 24 months, with total duration of study 4 years. Patients may discontinue from this NIS at any time.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the moment of ribociclib, alpelisib, monoET or CT treatment initiation.
2. Female gender.
3. Confirmed diagnosis of locally advanced/metastatic not amenable to surgery HR+/HER2- BC (progressed following prior therapy or de novo) for whom the treating physicial took the decision to initiate treatment with ribociclib, alpelisib, monoET or CT before entering the study.
4. Patient who initiated treatment with ribociclib, alpelisib, monoET or CT no longer than 4 weeks (28 days) prior to written informed consent for this study.
5. Patients with ECOG performance status ≤ 2.
6. Provision of written informed consent.

Exclusion Criteria:

1. Patients with a life expectancy of less than 3 months at the time of aBC diagnosis per the investigator's judgment.
2. Patients participating in any interventional clinical trial that includes investigational or marketed products at the time of enrollment. (Patients participating in other investigator initiated trial or NIS can be included as long as their standard of care is not altered by the study).
3. Patients receiving active treatment for malignancies other than BC at the time of enrollment.
4. Patients who are unable to understand the nature of the study.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with HR+/ HER2- advanced or metastatic BC that initiated treatment with ribociclib, alpelisib, monoET or CT within the study enrollment timeline
Study Population: Women with HR+/ HER2- advanced or metastatic BC that initiated treatment with ribociclib, alpelisib, monoET or CT within the study enrollment timeline will be provided by national oncology centers and hospitals that will be selected based on their experience in treating Breast Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2424 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) | Up to 24 months
  Defined as the time from study treatment initiation to the earliest of date of progression, date of death due to any cause, or date of discontinuation due to reasons other than 'Protocol violation' or 'Administrative problems'. The time to treatment failure for patients who did not experience treatment failure will be censored at last adequate tumor assessment.

SECONDARY OUTCOMES:
Line of treatment | Baseline
  Line of advanced breast cancer therapy when treatment of interest was prescribed
  * 1st
  * 2nd
  * 3rd
  * Later lines
ECOG status | Up to 24 months
  Eastern Cooperative Oncology Group (ECOG) Performance status: describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). Scores can range from a lower value of 0 (fully active, able to carry on all pre-disease performance without restriction) up to 5 (dead)
Location of metastases | Baseline
  Locations of metastatic sited at study entry:
  * Local
  * Lung
  * Liver
  * Central nervous system (CNS)
  * Bone
  * Other
Menopausal status | Baseline
  Menopausal status
  * Premenopausal
    * Ovarian suppression
    * Ovarian ablation
  * Perimenopausal
    * Ovarian suppression
    * Ovarian ablation
  * Postmenopausal
Number of patients with comorbidities | Baseline
  Number of patients with comorbidities will be presented
PIK3CA mutation status | Baseline
  PIK3CA mutation status
  * Confirmed PIK3CA mutation
  * Confirmed absence of PIK3CA mutation
  * No data available
Proportions of patients by treatment pattern | Up to 24 months
  Proportions of patients receiving the pre-stablished treatments
Proportions (%) of patients by treatment sequence | Up to 24 months
  Proportions (%) of patients by treatment sequence:
  * ribociclib in 1st line --> alpelisib in 2nd line.
  * alpelisib in 1st line --> ribociclib or other CDK4/6 inhibitor in 2nd line
Progression free survival (PFS) | Up to 24 months
  Defined as the time from index date to the date of the first documented progression or death due to any cause. If a patient has not had an event, PFS will be censored at the date of the last adequate tumor assessment by local BC management guidelines.
Overall survival (OS) | Up to 24 months
  Defined as the time from index date to date of death due to any cause. If a patient is not known to have died, then OS will be censored at the latest date the patient was known to be alive (on or before the cut-off date).
Time to chemotherapy (TTC) | Up to 24 months
  Defined as the time from index date to the date of initiation of chemotherapy in patient who did not receive chemotherapy for advanced breast cancer at the inclusion. The time to chemotherapy for patients who did not receive any chemotherapy will be censored at the end of follow-up period.
Proportion (%) of patients with permanent discontinuation | Up to 24 months
  Proportion of patients with permanent discontinuation to becollected
Reasons of permanent discontinuation | Up to 24 months
  Reason of treatment discontinuation (if initial treatment was discontinued)
  * Cancer progression
  * Adverse event
  * Death
  * Patient decision
  * Other
Proportion (%) of patients with dose adjustment | Up to 24 months
  Proportion of patients with dose adjustment will be collected
Reasons of dose adjustment | Up to 24 months
  Reasons of dose adjustment will be collected
Quality of life (EORTC QLQ-C30) | Baseline
  The changes from baseline to each visit where measured using QLQ-C30. EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Subject's responses to 28 questions about their physical functioning, disease symptoms, global health status and utilities are scored on a 4-point scale (1=Not at all to 4=Very much), a low score indicates a high / healthy level of functioning. And the responses to 2 questions about health-related QoL are scored on a 7-point scale (1=Very poor to 7=Excellent), a high score indicates a high / healthy level of functioning.
  Using linear transformation, raw scores are standardized, so that scores range from 0 to 100.
Quality of life (EQ-5D-5L) | Baseline
  EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3=moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (50):
- Russia (50):
  - Novartis Investigative Site, Syktyvkar, Komi
  - Novartis Investigative Site, Sochi, Russian Federation
  - Novartis Investigative Site, Kaluga, Russia
  - Novartis Investigative Site, Surgut, Tymen Area
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Belgorod
  - Novartis Investigative Site, Bryansk
  - Novartis Investigative Site, Cheboksary
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Cherkessk
  - Novartis Investigative Site, Chita
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Ivanovo
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kaliningrad
  - Novartis Investigative Site, Khabarovsk
  - Novartis Investigative Site, Khanty-Mansiysk
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Kostroma
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Moscow Region Balas
  - Novartis Investigative Site, Nal'chik
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Odintsovo
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Podolsk
  - Novartis Investigative Site, Pyatigorsk
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saransk
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Sevastopol’
  - Novartis Investigative Site, Severodvinsk
  - Novartis Investigative Site, Simferopol
  - Novartis Investigative Site, Tambov
  - Novartis Investigative Site, Tula
  - Novartis Investigative Site, Tver'
  - Novartis Investigative Site, Tyumen
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Vladikavkaz
  - Novartis Investigative Site, Vladivostok
  - Novartis Investigative Site, Voronezh
  - Novartis Investigative Site, Yekaterinburg
  - Novartis Investigative Site, Yuzhno-Sakhalinsk

IPD SHARING:
Plan to Share IPD: No